CLINICAL TRIAL: NCT00429572
Title: Mini-Allogeneic Peripheral Blood Progenitor Cell Transplantation For Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM97-268
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Results first posted 2011-07-13 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; PBPC Transplantation; Stem Cell Infusion; Fludarabine; Melphalan
MeSH Terms: conditions — Breast Neoplasms | interventions — fludarabine; Melphalan; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Allogeneic Transplantation (Experimental): Intravenous Fludarabine 30 mg/m^2 daily on days 1-5, and Melphalan 70 mg/m^2 on days 4 and 5 followed by blood stem cell transplant on day 7.
  Interventions: Drug: Fludarabine; Drug: Melphalan; Procedure: Stem Cell Infusion

INTERVENTIONS:
Drug: Fludarabine — 30 mg/m^2 intravenously Daily for 5 Days
Drug: Melphalan — 70 mg/m^2 intravenously Daily for 2 Days
Procedure: Stem Cell Infusion — Stem Cell Infusion on Day 0.
  Other Names: mini-allogeneic PBPC transplantation; Stem Cell Transplant; SCT

SUMMARY:
Primary Objectives:

1. To assess the feasibility of mini-allogeneic Peripheral Blood Progenitor Cell (PBPC) transplantation in patients with recurrent or metastatic breast cancer.
2. To determine the success rate (complete remission without severe toxicity or death) at 100 days after the transplant and long-term progression free survival (PFS) rate.
3. To examine the graft vs. breast cancer effect of allogeneic PBPC transplantation.

DETAILED DESCRIPTION:
If tumors shrink by standard-dose chemotherapy, patients will receive moderate dose chemotherapy to prepare for the blood stem cell transplant. The drug fludarabine will be given by vein on days 1-5. The drug melphalan will be given by vein on days 4 and 5. Day 6 will be a rest day; no drugs will be given. The blood stem cell transplant will be given on day 7. Bone marrow from the matched donor may be used instead of blood stem cells, particularly for unrelated donors. A catheter (tube) will be placed in a large vein in the chest to reduce the number of times patients are stuck with a needle.

Researchers will collect blood stem cells from your brother or sister or from an unrelated donor using granulocyte colony-stimulating factor (G-CSF) before receiving high-dose chemotherapy. You will need to have enough stem cells before transplantation.

The drugs G-CSG, tacrolimus, and methotrexate will be given to ease side effects and help blood counts return to normal after the transplant. G-CSF is given as a shot under the skin, starting the day from transplant and continuing until the white blood cell count is normal. Tacrolimus is given by vein or by mouth for 4 to 7 months; during the last month it is given, the dose will be tapered off. Methotrexate is given by vein on days 1, 3, and 6 after transplant. Day 11 of methotrexate is given additionally if a donor is unrelated. Blood transfusions may be needed also.

Antithymocyte globulin will be given to patients who receive blood or bone marrow from donors whose cells do exactly match the patients or from unrelated donors.

Sometimes the transplanted cells attack the normal cells in the patient's body instead of the cancer cells. This is called graft-vs-host disease (GVHD). The drug methylprednisolone will be given by vein or by mouth to fight GVHD is it occurs.

Patients must stay in the hospital for about 3 to 4 weeks. Patients must stay in the Houston area for about 100 days after the transplant. Blood tests will be done daily while the patient is in the hospital. Blood and urine tests and chest x-rays, computer tomography (CT) scans, and/or bone scans will be done during the 100 days.

If there are no signs of disease after 100 days, treatment will stop. Patients must return to the clinic for check-ups once a month for the first year, 3 times a year for 4 years, and once a year after that. If disease is till present after 100 days, but the patient does not have GVHD, the patient may receive an infusion of donor lymphocytes by vein. This treatment may be repeated up to 3 times with 8 weeks between infusions. If no disease is found or if GVHD occurs, treatment will stop.

Before treatment starts, patients will have a complete exam including blood and urine tests. An EKG (heart function test) and a heart scan will be done. Patients will have a dental exam. A test of lung function will be done. A sample of breast tissue will be taken. This is done with a hollow needle while the doctor looks at a CT scan or with a lighted tube placed through a cut in the breast while the patient is under anesthesia.

Herceptin will be given every week, if you have Human Epidermal growth factor Receptor 2 (HER-2)/neu-overexpressing tumor. Prior to this an infusion heart test will be done.

This is an investigational study. Docetaxel, Melphalan, and Herceptin are approved by the US Food and Drug Administration for use against breast cancer. About 40 patients will take part in the study.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or residual metastatic breast carcinoma
* Zubrod performance status less than 2
* 18-60 years old
* Related donor human leukocyte antigen (HLA)-compatible for allogeneic transplantation or unrelated HLA-compatible donor.
* No major organ dysfunction or active infection

Exclusion Criteria: None

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 1998-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoto Ueno, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period of January 1999 to December 2006. All participants were recruited at University of Texas MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Allogeneic Transplantation
Started | 19
Completed | 18
Not Completed | 1
Not completed — Disease progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Allogeneic Transplantation
Number analyzed (Participants) | 19
Age Continuous [Median (Full Range); unit: years] | 41 [31 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 19
Tumor Characteristic [Number; unit: participants] — Stage and Biomarkers
  participants
    ER negative | 12
    ER positive | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Tumor Response
Description: Best response recorded from start of treatment until disease progression/recurrence using World Health Organization (WHO) criteria of Complete Response: disappearance of all disease/symptoms > 4 weeks; Partial response, > 50% reduction in sum of products of diameters of each measurable lesion for more than 4 weeks; Stable Disease, no change in tumor size; and Progressive Disease, appearance of new lesions or > 25% increase in sum of products of diameters of any measurable lesions.
Time Frame: Baseline to measured progressive disease (post study follow-up period 24 months starting from the date of the last drug administration). Data collected every 4 months.
Population: As treated: Eighteen received the allogeneic transplantation.
Measure: Number; unit: participants
Arm/Group | Allogeneic Transplantation
Number analyzed (Participants) | 18
participants
  Complete Response | 5
  Stable Disease | 9
  Partial Response | 1
  Progressive Disease | 3

2. Primary Outcome: Overall Survival
Description: Survival duration was calculated from time of transplantation by number of days.
Time Frame: Transplant until death.
Population: As treated: Eighteen received the allogeneic transplantation.
Measure: Median (Full Range); unit: Days
Arm/Group | Allogeneic Transplantation
Number analyzed (Participants) | 18
Days | 643 [57 to 2526]

3. Primary Outcome: Time to Progressive Disease
Description: Progression-free was measured, by days, at time from transplantation to development to disease or death from any cause, which ever occurred first.
Time Frame: Transplant to Progression.
Measure: Median (Full Range); unit: Days
Arm/Group | Allogeneic Transplantation
Number analyzed (Participants) | 18
Days | 202 [43 to 1063]

4. Primary Outcome: Grade II-IV Toxicity
Description: Non-hematopoietic toxicity within the first year of transplantation, acute Graft versus Host Disease (GVHD) above National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade I and chronic above Grade I are reported by participant incidence. Broad classification of adverse events (AE) categories based on anatomy and/or pathophysiology; within each category, AEs are listed accompanied by their descriptions of severity (Grade, Grade 1 least severe).
Time Frame: Up to one year.
Population: As treated: Eighteen received the allogeneic transplantation.
Measure: Number; unit: Participants
Arm/Group | Allogeneic Transplantation
Number analyzed (Participants) | 18
Participants
  Cardiac | 1
  Pulmonary | 3
  Gastrointestinal | 8
  Renal | 0
  Neurological | 2
  Fever/Flu like symptoms | 2
  Infection | 3
  Genitourinary | 2
  Skin | 2

5. Primary Outcome: Number of Participants With Acute or Chronic GVHD And Response to Therapy
Description: Participants diagnosed with Graft versus Host Disease (GVHD) post transplant were divided into either acute (aGVHD), normally observed within the first 100 days post-transplant; and chronic GVHD (cGVHD) cases, normally occur after 100 days, then evaluated and scored according to standard criteria from "Consensus conference on acute GVHD grading," Bone Marrow Transplant 1995; 15: 825-828, noted is type of case and whether responds to therapy.
Time Frame: Transplant to 1 year post transplant
Population: As treated: Eighteen received the allogeneic transplantation.
Measure: Number; unit: participants
Arm/Group | Allogeneic Transplantation
Number analyzed (Participants) | 18
participants
  aGVHD | 9
  aGVHD responded to therapy | 7
  cGVHD | 14
  cGVHD responded to therapy | 14

ADVERSE EVENTS:
Time Frame: 7 Years
Description: Cardiac 1 Pulmonary 3 Gastrointestinal 8 Renal 0 Neurological 2 Fever/Flu like symptoms 2 Infection 3 Genitourinary 2 Skin 2
Arm/Group | Allogeneic Transplantation
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 9/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Allogeneic Transplantation (N=19)
Diarhhea (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 9
Vomitting (Gastrointestinal disorders) | 9
Skin rash (Skin and subcutaneous tissue disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No